CLINICAL TRIAL: NCT02498977
Title: Prospective Randomised Marker-based Trial to Assess the Clinical Utility and Safety of Biomarker-guided Immunosuppression Withdrawal in Liver Transplantation
Brief Title: Liver Immunosuppression Free Trial
Acronym: LIFT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary endpoint not reached.
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ASF/001-01; 2014-004557-14 (EudraCT Number)
Record Dates: First submitted 2015-06-11; First posted 2015-07-15 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Transplantation, Liver
Keywords: Liver; Transplant; Immunosuppression
MeSH Terms: interventions — Biomarkers; Tacrolimus; Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (weaning) (Active Comparator): All participants satisfying clinical criteria will be weaned off immunosuppression drugs irrespective of biomarker result.
  Interventions: Drug: Tacrolimus, cyclosporine and/or mycophenolic acid, mycophenolate mofetil or azathioprine
- Arm B+ (weaning- positive biomarker) (Active Comparator): Participants with a positive biomarker will be weaned of immunosuppression drugs.
  Interventions: Genetic: Biomarker
- Arm B- (maintenance) (Active Comparator): Participant with negative biomarker test result will be informed of the result and will remain on baseline maintenance immunosuppression drugs.
  Interventions: Genetic: Biomarker

INTERVENTIONS:
Genetic: Biomarker — Real time polymerase chain reaction (PCR) gene expression measurement
  Arms: Arm B+ (weaning- positive biomarker); Arm B- (maintenance)
Drug: Tacrolimus, cyclosporine and/or mycophenolic acid, mycophenolate mofetil or azathioprine — Immunosuppression drugs as per protocol
  Other Names: IS
  Arms: Arm A (weaning)

SUMMARY:
LIFT is prospective randomised marker-based trial to assess the clinical utility and safety of biomarker-guided immunosuppression withdrawal in liver transplantation. 'LIFT' aims to validate a biomarker test of operational tolerance to stratify liver transplant recipients before withdrawing immunosuppressive medication. Primary objective is clinical utility and risk/benefit ratio of employing a transcriptional test of tolerance to stratify liver recipients prior to immunosuppression withdrawal. Secondary objectives are: safety of biomarker-guided immunosuppression withdrawal; health-economic and quality of life impact of biomarker-guided immunosuppression withdrawal; improvement in drug-related co-morbidities; prevalence of tolerance over time; role of donor-specific anti-human leukocyte antigen (HLA) antibodies; identify mechanisms of liver allograft tolerance. It is a prospective, multi-centre, phase IV, biomarker-strategy design trial with a randomized control group in which adult liver transplant recipients will undergo immunosuppression withdrawal. The sample size is 148 patients.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, phase IV, biomarker-strategy design trial with a randomised control group in which adult liver transplant recipients will undergo immunosuppression (IS) withdrawal. Immunosuppression drugs (IS) are: Tacrolimus, cyclosporine and/or mycophenolic acid, mycophenolate mofetil or azathioprine.

Enrolled participants will be randomised 1:1 to either: 1) Non-Biomarker-based IS weaning (Weaning-All; Arm A); or 2) Biomarker-based IS weaning (Arm B). In participants allocated to Arm A IS will be withdrawn regardless of the result of the biomarker test. Among participants allocated to Arm B, only those found to be biomarker-positive (Arm B+, i.e. potentially tolerant) will be offered IS withdrawal, while biomarker-negative participants (Arm B-, i.e. potentially non-tolerant) will remain on their baseline maintenance IS. This will allow us to demonstrate that the biomarker is a useful test to personalise IS by offering drug withdrawal only to those participants who are likely to complete the process successfully, avoiding unnecessary rejections among those who have not developed tolerance. Comparing the outcome of IS withdrawal between arms A and B+ will provide direct evidence of the clinical usefulness of the test as a function of its predictive accuracy. We have established that for the biomarker to drive safe IS withdrawal its Positive Predictive Value should be no less than 0.80, and its sensitivity at least 070. To account for centre effects, we will use stratified randomization. Furthermore, to avoid biases, participants undergoing drug withdrawal and their physicians will be blinded to the biomarker results. Participants randomized to Arm B- will know their biomarker status, and will be maintained in the study until its termination and contribute to secondary clinical outcomes and to the evaluation of the stability of the tolerance signature.

Cost and quality of life (HrQOL) assessments will be conducted alongside the trial to estimate the health-economic implications of the 2 different strategies. Furthermore, sequential biological specimens will be collected to conduct ancillary mechanistic studies. Recruitment will take place in 11 European liver transplant units (King's College Hospital, Royal Free London, Newcastle, Birmingham, Leeds, Edinburgh, Cambridge, Leuven, Hannover, Berlin and Barcelona).

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening: more than 3 years post-transplant if participants are ≥50 years old, OR more than 6 years post-transplant if participant age is 18-49 years old.
2. Recipient of either deceased or living donor liver transplant.
3. Recipient of single organ transplant only
4. Liver function tests: direct bilirubin ≤17.1 umol/L and Alanine aminotransferase (ALT) ≤60 IU/L at the screening visit.
5. On calcineurin inhibitor (CNI) based maintenance IS and no more than one of the following: Low dose mycophenolic acid (≤ 1080 mg daily), mycophenolate mofetil (MMF ≤ 1500 mg daily), or azathioprine (≤ 150 mg daily); or on mycophenolate/mycophenolic monotherapy (effective contraception must be used before beginning mycophenolate therapy, during therapy, and for six weeks following discontinuation of therapy).
6. Ability to sign informed consent.

Exclusion Criteria:

1. Serum positivity for Hepatitis C virus (HCV-RNA)
2. Serum positivity for HIV-1 infection, Hepatitis B virus (HBV) surface antigen or HBV-DNA
3. Immune-mediated liver disease in which IS discontinuation is inadvisable (autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cirrhosis).
4. Acute or chronic rejection within the 52 weeks prior to screening.
5. Glomerular filtration rate (GFR) <40 mL/min (to mitigate the risk of worsening renal failure should rejection occur and high level of CNI be required).
6. The need for chronic anti-coagulation that cannot be safely discontinued to safely perform for a liver biopsy.
7. Baseline (screening) liver biopsy showing any of the following: a) acute rejection according to Banff criteria; b) early or late chronic rejection according to Banff criteria; c) inflammatory activity and/or fibrosis in excess of permissive criteria; f) any other findings that might make participation in the trial unsafe. Eligibility will be determined by the central pathologist.
8. Patient age <18 years old at the time of transplant.
9. Pregnant females and females of childbearing age not using effective contraception.
10. Current illicit drug or alcohol abuse.
11. Inability to participate in frequent monitoring of liver function (every 3 weeks) and clinical visits during IS withdrawal.
12. Inability to comply with study directed treatment.
13. Any medical condition that in the opinion of the principal investigator would interfere with safe completion of the trial.
14. Participation in another clinical trial during the month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Successful discontinuation of IS with maintenance of normal allograft status | 12 months from IS withdrawal
  Number of patients with successful discontinuation of IS with maintenance of normal allograft status as assessed by liver biopsy and liver tests 12 months after IS withdrawal (operational tolerance)

SECONDARY OUTCOMES:
Proportion of tolerant participants remaining free of rejection | 3 years post IS withdrawal
  Measures of rejection in patients (incidence, severity, timing, steroid resistant rejection, chronic rejection) and to investigate if liver transplant recipients under IS become operationally tolerant over time.
Renal function at 1, 2 and 3 years after enrollment and change in co-morbidities | 3 years post IS withdrawal
  To determine the extent to which IS withdrawal improve drug-related co-morbidities associated with IS use (hypertension, cardiovascular risk profile, diabetes mellitus, hyperlipidemia, malignancy) and to explore the association between operational liver transplant tolerance, iron metabolism, immunosenescence, and specific gut microbiome profiles.
Development of anti-HLA antibodies (before and after initiation of IS withdrawal). | 3 years post IS withdrawal
  To determine if the presence of donor-specific anti-HLA antibodies influence the success of IS withdrawal, and whether IS withdrawal promotes the development of anti-HLA antibodies in liver transplant recipients.
Change in Health related quality of life (HrQOL) | 3 years post IS withdrawal
  To assess the effect of IS withdrawal on the quality of life of liver transplant recipients.
Costs of treatment | 3 years post IS withdrawal
  Measuring pharmacoeconomic impact of IS withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle